CLINICAL TRIAL: NCT03424629
Title: A Randomized, Positive Controlled Trial That Assess the Safety And Efficacy of Umbilical Cord-Derived Mesenchymal Stem Cells in Moderate and Severe Plaque Psoriasis Patients
Brief Title: Safety and Efficacy of UC-MSCs in Patients With Plaque Psoriasis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Ever Union Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TianjinEverUnion
Record Dates: First submitted 2017-12-27; First posted 2018-02-07 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2017-12

CONDITIONS: Moderate and Severe Plaque Psoriasis
Keywords: psoriasis; UC-MSCs
MeSH Terms: conditions — Lymphoma, Follicular; Psoriasis | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Dose UC-MSCs (Experimental): Umbilical Cord Mesenchymal Stem Cells (UC-MSCs) 1 x 10^6 cells/kg in normal saline injection
  Interventions: Biological: Low-dose UC-MSCs
- High-Dose UC-MSCs (Experimental): Umbilical Cord Mesenchymal Stem Cells (UC-MSCs) 3 x 10^6 cells/kg in normal saline injection
  Interventions: Biological: High-dose UC-MSCs
- Methotrexate (Active Comparator): 5-25mg Methotrexate orally
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Biological: Low-dose UC-MSCs — Participants will receive 6 times UC-MSCs infusions (each time 1×10^6/kg). The first time to fourth time will be given once a week for successive 4 weeks（week 0,1,2,3）, then the last two times will be given once every two weeks（week 5,7）.
  Other Names: regenskin
  Arms: Low-Dose UC-MSCs
Biological: High-dose UC-MSCs — Participants will receive 6 times UC-MSCs infusions (each time 3×10^6/kg). The first time to fourth time will be given once a week for successive 4 weeks（week 0,1,2,3）, then the last two times will be given once every two weeks（week 5,7）.
  Other Names: regenskin
  Arms: High-Dose UC-MSCs
Drug: Methotrexate — Participants will be administered Methotrexate (each time 5-25mg) orally once a week for successive 16 weeks(week 0-15).
  Arms: Methotrexate

SUMMARY:
This is a study in patients with moderate to severe chronic plaque psoriasis.All the participants will be randomized into three groups, high-dose UC-MSCs, low-dose UC-MSCs, or methotrexate group.This study is designed to prove that UC-MSCs is safe and effective.

DETAILED DESCRIPTION:
Psoriasis is a chronic, incurable, immune-mediated dermatological disease, and it is considered that immune system dysregulation is the important cause of the disease.Umbilical cord derived mesenchymal stem cells (UC-MSCs) have be proven safe and effective for the treatment of various intractable autoimmune and inflammatory disorders because of their distinct immunomodulatory properties.

Patients will be randomized into three groups.In one group patients will be treated with 1x10^6 cells/kg in 0,1,2,3,5,7 week, in the second group patients will be treated with 3x10^6 cells/kg in 0,1,2,3,5,7 week,in the third group patients will be treated with 5-25mg Methotrexate from 0 to 15 week In this study, researchers will determine the safety of UC-MSCs that a patient can tolerate without causing side effects. Moreover researchers will also be assess the efficacy and sustainability of UC-MSCs in 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years old with moderate-to-severe psoriasis.
* Diagnosis of plaque psoriasis at least 6 months before entering the study.
* Moderate-to-severe plaque psoriasis(PASI≥10，or BSA≥10% and DLQI score≥10).
* Failure after conventional therapy.
* No other treatment for psoriasis during the period of the trial.
* Willing and able to comply with all study requirements and provide informed consent.

Exclusion Criteria:

* Other types of psoriasis,such as pustular, erythrodermic and guttate psoriasis).
* Drug-induced psoriasis (i.e., new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium).
* Ongoing use of other psoriasis treatments.
* Ever use of any biologic drug directly targeting IL-17,IL-23,TNFa etc.
* Active systemic infections during the last two weeks (exception: common cold) prior to initiation of the trial and any infections that reoccur on a regular basis.
* History of malignancy .
* Evidence of infection with HIV, hepatitis B or hepatitis C.
* Pregnant or lactating females, or willing to have a baby during the trial.
* Can not be traced on time.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who have 75% or more reduction in [Psoriasis area-and-severity index score (PASI)] (PASI75) at week 20 | Week 20
  The proportion of subjects who have a reduction of 75% or more from baseline in the psoriasis area-and-severity index score (PASI 75) at week 20
Proportion of subjects who achieve a score of 0 or 1 on a 5-point Physician's global assessment（PGA0/1) at week 20 | Week 20
  The proportion of subjects who achieve a score of 0（clear）or 1（almost clear）on a 5-point Physician's global assessment（PGA0/1) at week 20

SECONDARY OUTCOMES:
Proportion of subjects who have 90% or more reduction in [Psoriasis area-and-severity index score (PASI)] (PASI90) at week 20 | Week 20
  The proportion of subjects who have a reduction of 90% or more from baseline in the psoriasis area-and-severity index score (PASI 90) at week 20
Proportion of subjects who have 75% or more reduction in [Psoriasis area-and-severity index score (PASI)] (PASI75) at week 12,16,36,52 | Week 12,16,36,52
  The proportion of subjects who have a reduction of 75% or more from baseline in the psoriasis area-and-severity index score (PASI 75) at week 12,16,36,52
Proportion of subjects who achieve a score of 0 or 1 on a 5-point Physician's global assessment（PGA0/1) at week 12,16,36,52 | Week 12,16,36,52
  The proportion of subjects who achieve a score of 0（clear）or 1（almost clear）on a 5-point Physician's global assessment（PGA0/1) at week 12,16,36,52
Frequency of Adverse Events and Serious Adverse Events | Week 0 through week 52
  Frequency of all Adverse Events (AEs) and Serious Adverse Events (SAEs) that occur during the whole trial including the observational period (AEs and SAEs include but not limited to headaches, allergies, fever and so on
Proportion of subjects who experience psoriasis relapse | Week 8 though week 52
  The proportion of subjects who experience a psoriasis relapse at any time until week 52. Psoriasis relapse is defined as loss of > 50% of the initial PASI improvement measured at week 7

OTHER OUTCOMES:
Change from Baseline in Dermatology Life Quality Index (DLQI) score though 52 weeks | Week 0,1,2,3,5,7,12,16,20,36,52
  DLQI score will be assessed at week 0,1,2,3,5,7,12,16,20,36,52
Exploring the theoretical basis of stem cell therapy for psoriasis | 0,1,2,3,5,7 12,16,20,36,52 week
  Analysis the serum cytokine content, immunological subgroup and pathological section to explore the theoretical basis of stem cell therapy for psoriasis

CONTACTS AND LOCATIONS:
Overall Officials: Chunlei Zhang, doctor, Study Chair — Peking University Third Hospital; Xin Guan, doctor, Principal Investigator — Peking University Third Hospital; Chunting Li, doctor, Principal Investigator — Peking University Third Hospital; Jinzhu Guo, doctor, Principal Investigator — Peking University Third Hospital; Wenhui Wang, doctor, Study Director — Peking University Third Hospital
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing
  - Tianjin Ever Union Biotechnology Co., Ltd., Beijing

IPD SHARING:
Plan to Share IPD: No